CLINICAL TRIAL: NCT00879853
Title: Randomized Controlled Trial of Mental Health Treatment for Darfur Refugees in Cairo
Brief Title: Trial of Mental Health Treatment for Darfur Refugees in Cairo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Ma'an Organization (Other)
Responsible Party: Charles Marmar, M.D., University of California, San Francisco
Other Study IDs: UCSF Academic Senate Grant
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Post-Traumatic Stress Disorder; Depression; Anger; Domestic Violence
Keywords: PTSD; Depression; Anger; Domestic Violence; Refugee; Asylum Seeker; Community Therapist; Paraprofessional Therapists
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpersonal Therapy (Experimental)
  Interventions: Behavioral: Interpersonal Therapy
- Wait List Control (No Intervention)

INTERVENTIONS:
Behavioral: Interpersonal Therapy
  Arms: Interpersonal Therapy

SUMMARY:
The enormous global burden of mental illness has been estimated through the publication of the Global Burden of Disease Study, adding momentum to refugee mental health studies (1,2). As research confirms that high levels of Posttraumatic Stress Disorder (PTSD) and depression occur in post-conflict settings, it is essential to develop effective treatment for psychological trauma in refugee populations recovering from mass violence (3-4). PTSD and depression are risk factors for anger, interpersonal discord and violence, not only among those who have trauma and depression, but also among their spouses and children (5-9). This "infectious" model of trauma/violence is critically important in the setting of ethnic conflict, as increased levels of interpersonal violence within the afflicted community hinder its recovery and fuel future cycles of conflict. To date, there has been little research on the interpersonal effects of trauma among refugee populations. The proposed research is a pilot and randomized controlled trial of "Interpersonal Therapy" (IPT) for Sudanese refugees living in Cairo. IPT, a very effective therapy for depression, has been adapted for PTSD treatment and sub-Saharan Africa settings (10-12). Measures will evaluate success of the treatment not only in terms of individual PTSD and depression symptoms, but also with respect to interpersonal conflict. Hypotheses: (1) After IPT intervention, Sudanese refugees will have lower levels of depression and trauma symptoms compared to wait list controls (2) After IPT intervention, Sudanese refugees will have lower levels of interpersonal violence compared to wait list controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years;
2. Absence of cognitive dysfunction which requires a higher level of care and/or interferes with ability to participate in IPT;
3. Absence of severe thought or mood disorder symptoms which requires a higher level of care and/or interferes with ability to participate in IPT;
4. Absence of drug and alcohol dependence;
5. HTQ score of 2.3 or greater;
6. Ability to attend twice a week therapy sessions for 4 weeks and return for regular screening;
7. Ability to give verbal informed consent .

Exclusion Criteria:

1. Unable to give informed consent;
2. Age less than 18;
3. Cognitive dysfunction which requires a higher level of care and/or interferes with ability to participate in IPT;
4. Severe thought or mood disorder symptoms which requires a higher level of care and/or interferes with ability to participate in IPT;
5. Drug or alcohol dependence in the past 6 months;
6. HTQ score less than 2.5;
7. Inability to attend twice a week therapy sessions for 4 weeks and return for regular screening .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder Symptoms

SECONDARY OUTCOMES:
Depression Symptoms
Anger
Household Conflict/Violence

CONTACTS AND LOCATIONS:
Locations (1):
- Ma'an Organization, Cairo, Egypt